CLINICAL TRIAL: NCT02819011
Title: OHI--Randomized Control Trial to Evaluate Efficacy, Acceptability, and Perception of Benefit of an Innovative Custom AFO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bijan Najafi, PhD (Other)
Collaborators: Orthotic Holdings, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-38050
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Accidental Falls; Fall Due to Loss of Equilibrium; High Risk of Falls Due to Mobility Limitation; Diabetes; Arthritis; Cancer; Peripheral Arterial Disease; Parkinson's Disease; End Stage Renal Failure on Dialysis
Keywords: Ankle Foot Orthoses; falls; Fall Prevention; Frailty; Concern for falls; Footwear; Mobility
MeSH Terms: conditions — Diabetes Mellitus; Arthritis; Neoplasms; Peripheral Arterial Disease; Parkinson Disease; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBB AFO Group (Experimental): This group will be provided with a pair of New Balance 813 shoes plus a custom made MBB AFO for the duration of the study.
  Interventions: Device: MBB AFO
- No MBB AFO Group (Active Comparator): This group will be provided with a pair of New Balance 813 shoes for the duration of the study.
  Interventions: Other: Control

INTERVENTIONS:
Device: MBB AFO — Subjects will be provided with a pair of New Balance 813 shoes plus a custom made MBB AFO
  Arms: MBB AFO Group
Other: Control — Subjects will be provided with a pair of New Balance 813 shoes
  Arms: No MBB AFO Group

SUMMARY:
The investigators propose a randomized control trial to evaluate long term effects and effectiveness of Moore Balance Brace (MBB) ankle foot orthoses (AFO) in reducing risk of falling in older adults.

Primary Endpoints • Characterize the impact of MBB AFO on balance, gait, risk of falling, frailty status, and adverse events

Secondary Endpoints • Characterize the Impact of MBB AFO on spontaneous daily physical activities • Characterize the feasibility of the MBB AFO device on patient adherence, acceptability, user-friendliness, and perception of benefit for daily usage

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* High concerns or high risk of fall
* Ambulatory

Exclusion Criteria:

* Presence of an active wound infection on either of the foot and ankle
* Use of medication or a medical condition that may have unstable (fluctuate over time) or temporary (less than one month) impact on gait and balance
* Acute fractures on the foot
* Participant of an interventional study within the last 30 days
* Non-ambulatory or unable to stand without help or walk a distance of at least 1.8 m (~six feet) without assistance
* Major foot amputation
* Unable or unwilling to participate in all procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only de-identified data and associated results will be published in peer-reviewed papers or scientific abstracts

REFERENCES:
- [Result] Wang C, Goel R, Rahemi H, Zhang Q, Lepow B, Najafi B. Effectiveness of Daily Use of Bilateral Custom-Made Ankle-Foot Orthoses on Balance, Fear of Falling, and Physical Activity in Older Adults: A Randomized Controlled Trial. Gerontology. 2019;65(3):299-307. doi: 10.1159/000494114. Epub 2018 Nov 30. PMID 30504728
- [Result] Wang C, Goel R, Zhang Q, Lepow B, Najafi B. Daily Use of Bilateral Custom-Made Ankle-Foot Orthoses for Fall Prevention in Older Adults: A Randomized Controlled Trial. J Am Geriatr Soc. 2019 Aug;67(8):1656-1661. doi: 10.1111/jgs.15929. Epub 2019 Apr 24. PMID 31018018

RESULTS

PARTICIPANT FLOW:
Groups:
- Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group: This group will be provided with a pair of New Balance 813 shoes plus a custom made Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) for the duration of the study.
  Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO): Subjects will be provided with a pair of New Balance 813 shoes plus a custom made Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO)
- No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group: This group will be provided with a pair of New Balance 813 shoes for the duration of the study.
  Control: Subjects will be provided with a pair of New Balance 813 shoes
Period: Overall Study
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Started | 22 | 22
Completed | 15 | 17
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (6.3) | 75.6 (6.5) | 74.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Hip Sway Change From Baseline to 6 Months
Description: Hip sway (motion of hip joints in three dimensions) measured by wearable sensors while wearing their own shoes compared to the orthopedic shoes and compared to orthopedic shoes plus Ankle-Foot Orthosis (AFO)
Time Frame: baseline to 6 months
Population: Some participants in AFO and No AFO groups withdrew from study in 6 months. Mixed Model Analysis can handle such missing data
Measure: Mean (Standard Deviation); unit: degree^2
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
degree^2
  Baseline | 3.65 (3.22) | 3.75 (3.63)
  @6Month: number analyzed (Participants) | 14 | 18
  @6Month | 2.15 (1.24) | 3.89 (2.15)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare changes in two groups from baseline to 6 months; Test type: Superiority; p = 0.040, Mixed Models Analysis — priori threshold for statistical significance= 0.05

2. Primary Outcome: Ankle Sway Change From Baseline to 6 Months
Description: Ankle sway (motion of ankle joint in three dimensions) measured by wearable inertial sensors while wearing their own shoes compared to the orthopedic shoes and compared to orthopedic shoes plus Ankle-Foot Orthosis (AFO)
Time Frame: baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree^2
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
degree^2
  Baseline | 3.50 (3.74) | 3.21 (2.43)
  @6Month: number analyzed (Participants) | 14 | 18
  @6Month | 1.03 (0.69) | 3.56 (2.54)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes in both groups from baseline to 6 months; Test type: Superiority; p = 0.005, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

3. Primary Outcome: Center of Mass (COM) Sway Change Baseline to 6 Months
Description: Center of Mass (COM) sway measured by wearable inertial sensors while wearing their own shoes compared to the orthopedic shoes and compared to orthopedic shoes plus Ankle-Foot Orthosis (AFO)
Time Frame: baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
cm^2
  Baseline | 0.71 (0.50) | 0.85 (0.65)
  @6Month: number analyzed (Participants) | 14 | 18
  @6Month | 0.32 (0.18) | 0.76 (0.54)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes in both groups from baseline to 6 months; Test type: Superiority; p = 0.019, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

4. Secondary Outcome: Adherence (Hours Per Day to Wear Ankle-Foot Orthosis (AFO))
Description: The adherence of participants to the prescribed Ankle-Foot Orthosis (AFO) plus walking shoes was quantified using the response to a self-reported question ("How many hours per day did you wear the prescribed footwear?").
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 14 | 13
hours per day | 5.4 (3.3) | 5.6 (3.2)

5. Secondary Outcome: Fall Incidents
Description: Fall incidents during the study
Time Frame: Baseline, 12 months
Population: Some participants in AFO and No AFO groups withdrew from study in 6 and 12 months. Generalized Estimating Equation Analysis can handle such missing data
Measure: Mean (Standard Deviation); unit: falls per year precedent
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
falls per year precedent
  Baseline | 2.27 (4.17) | 1.82 (4.19)
  @12Month: number analyzed (Participants) | 15 | 14
  @12Month | 0.80 (1.27) | 0.94 (1.25)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes of both groups from pre-intervention to post-intervention year; Test type: Superiority; p = 0.572, Generalized Estimating Equations — priori threshold for statistical significance = 0.05

6. Secondary Outcome: Concern for Falling Change Form Baseline to 6 Months
Description: Concern for falling is quantified by Falls Efficacy Scale - International (FES-I) questionnaire. Scores range from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling). Higher score indicate worse performance.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group: This group will be provided with a pair of New Balance 813 shoes plus a custom made Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) for the duration of the study.
  Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) : Subjects will be provided with a pair of New Balance 813 shoes plus a custom made Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO)
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
score on a scale
  Baseline | 32.8 (10.7) | 33.3 (11.5)
  @6Month: number analyzed (Participants) | 14 | 18
  @6Month | 27.0 (9.0) | 30.1 (13.9)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes between groups from baseline to 6 months; Test type: Superiority; p = 0.650, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

7. Secondary Outcome: Physical Activity Level
Description: Physical activity level for 24 hours while wearing their own shoes compared to the walking shoes and compared to walking shoes plus Ankle-Foot Orthosis (AFO). To quantify physical activity, number of taken steps per day was monitored using a pendant wearable sensor called, PAMSys (Biosensics, MA, USA).
Time Frame: baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of steps per day
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
number of steps per day
  Baseline | 4017 (2008) | 3847 (3645)
  @6Month: number analyzed (Participants) | 14 | 18
  @6Month | 4872 (2657) | 4297 (2735)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes between groups from baseline to 6 months; Test type: Superiority; p = 0.756, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

8. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events reported during the study. Adverse events was inquired at 1 months, 3 months, 6 months, 12 months after the baseline, and summed at 12 months. If the participant has at least one adverse event reported in any assessed time frame, the participant will be categorized as the participant with adverse event.
Time Frame: assessed at 1, 3, 6, and 12 months, month 12 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

9. Secondary Outcome: Percentage of Participants Who Found the Device Useful and Easy to Use
Description: The participants perceived usefulness of ease of use of wearing Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) based on questionnaires of A technology acceptance model (TAM). Perceived usefulness was assessed using two questions (i.e., "I feel more stable when standing," and "I feel more stable when walking"). Perceived ease of use was assessed using two questions (i.e., "Was easy to take on and off," and "Was comfortable to wear"). The Likert scale (6-point scale from 0-5) was used to quantify how much they disagreed with each statement, including "strongly disagree," "disagree," "somewhat disagree," "somewhat agree," "agree," and "strongly agree," respectively. In this paper, responses were only categorized as positive (3-5 points) or negative (0-2 points) attitudes towards the use of AFO plus walking shoes.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 14
percentage of participants
  perceived usefulness | 79
  perceived ease of use | 93

10. Secondary Outcome: Stride Velocity
Description: stride velocity measured in single-task walking with normal speed
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
m/sec
  Baseline | 0.80 (0.23) | 0.81 (0.27)
  6 months: number analyzed (Participants) | 14 | 18
  6 months | 0.88 (0.27) | 0.88 (0.30)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes between groups from baseline to 6 months; Test type: Superiority; p = 0.769, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

11. Secondary Outcome: Stride Time
Description: stride time measured in single task walking with normal speed
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
seconds
  Baseline | 1.27 (0.18) | 1.24 (0.21)
  6 months: number analyzed (Participants) | 14 | 18
  6 months | 1.25 (0.23) | 1.21 (0.18)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes between groups from baseline to 6 months; Test type: Superiority; p = 0.857, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

12. Secondary Outcome: Stride Length
Description: stride length measured in single-task walking with normal speed
Time Frame: baseline, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
Number analyzed (Participants) | 22 | 22
meters
  Baseline | 0.98 (0.17) | 0.96 (0.22)
  6 months: number analyzed (Participants) | 14 | 18
  6 months | 1.05 (0.22) | 1.01 (0.27)
Statistical Analysis 1: Comparison: Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group vs No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group; Repeated measures to compare the changes between groups from baseline to 6 months; Test type: Superiority; p = 0.829, Mixed Models Analysis — a priori threshold for statistical significance = 0.05

ADVERSE EVENTS:
Time Frame: 1 year
Description: Incident of falls related to footwear/AFO, pain, and other relevant adverse events such as callus, foot ulcers, etc
Arm/Group | Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group | No Moore Balance Brace (MBB) Ankle-Foot Orthosis (AFO) Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT02819011/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT02819011/SAP_001.pdf